CLINICAL TRIAL: NCT05292521
Title: Utilizing Patient Reported Quality of Life to Inform Patient Decision Making in Early-Stage Lung Cancer
Brief Title: Quality of Life Intervention to Inform Patient Decision-Making in Early-Stage Lung Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Comprehensive Cancer Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: I 2220321; NCI-2022-01257 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 2220321 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2022-03-03; First posted 2022-03-23 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Lung Non-Small Cell Carcinoma; Stage I Lung Cancer AJCC v8; Stage IA1 Lung Cancer AJCC v8; Stage IA2 Lung Cancer AJCC v8; Stage IA3 Lung Cancer AJCC v8; Stage IB Lung Cancer AJCC v8; Stage II Lung Cancer AJCC v8; Stage IIA Lung Cancer AJCC v8; Stage IIB Lung Cancer AJCC v8
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Practice Guidelines as Topic; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (QOL fact sheet) (Experimental): Patients receive study QOL intervention fact sheet during the initial consult that occurs 4 weeks prior to the standard of care surgery or SBRT. Patients have an opportunity to review the QOL fact sheet in person and discuss any questions with the treating physician(s).
  Interventions: Other: Informational Intervention; Other: Questionnaire Administration
- Group B (usual care) (Active Comparator): Patients receive usual care during the initial consult that occurs 4 weeks prior to the standard of care surgery or SBRT.
  Interventions: Other: Best Practice; Other: Questionnaire Administration

INTERVENTIONS:
Other: Best Practice — Receive usual care
  Other Names: standard of care; standard therapy
  Arms: Group B (usual care)
Other: Informational Intervention — Receive QOL fact sheet
  Arms: Group A (QOL fact sheet)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This clinical trial studies the effect of a quality of life intervention on decision-making in patients with early-stage lung cancer who are undergoing standard of care surgery or stereotactic body radiation therapy (SBRT). Providing quality of life outcome data to patients deciding between surgery and SBRT may help decrease decision regret and increase patient satisfaction with their care.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine the effect of provision of quality-of-life (QOL) information versus usual care for standard of care surgery or SBRT treatment on decision regret.

SECONDARY OBJECTIVES:

I. Determine the effect of provision of QOL information versus usual care for standard of care surgery or SBRT treatment on QOL measures.

II. Determine the influence of socioeconomic status on the relationship between decision regret and QOL information associated with each treatment modality.

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP A: Patients receive study QOL intervention fact sheet during the initial consult that occurs 4 weeks prior to the standard of care surgery or SBRT. Patients have an opportunity to review the QOL fact sheet in person and discuss any questions with the treating physician(s).

GROUP B: Patients receive usual care during the initial consult that occurs 4 weeks prior to the standard of care surgery or SBRT.

Patients are followed up at 1, 3, and 6 months after standard of care surgery or SBRT.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Radiographic stage I-II non-small cell lung cancer (NSCLC)

  * Of note, separate tumor nodule(s) in an ipsilateral lobe different from that of the primary is considered T4 disease. However, these are treated as separate stage I or II lesions and will be eligible for this study.
* Eligible for both surgery and SBRT
* Able to provide informed consent in English
* Have verbal fluency in English
* Participant must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

* Radiographic stage III-IV NSCLC except as noted above
* Eligible for either only surgery or SBRT, but not both
* Eligible for palliative-intent treatments or supportive care only.
* Pregnant female participants.
* Unwilling or unable to follow protocol requirements
* Any condition which in the investigator's opinion deems the participant an unsuitable candidate
* Cognitively impaired adults/adults with impaired decision-making capacity
* Individuals who are not yet adults (infants, children, teenagers)
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-12-21 (Actual); Primary Completion 2028-12-21 (Estimated); Study Completion 2028-12-21 (Estimated)

PRIMARY OUTCOMES:
Decision regret | At 6 months
  Compare the extent of decision regret based on Decision Regret Scale between the provision of quality of life (QOL) information versus usual care for standard of care surgery or stereotactic body radiation therapy (SBRT) treatment. The five-point decision regret score will be converted to a 100-point score as described by others, where a higher score reflects an increased decision regret. In this schema, a decision regret score > 25 % is deemed moderate to severe regret. The dichotomized decision regret will be modeled as a function of group, time, and their interaction using a generalized estimating equations (GEE) logistic regression model with an autoregressive covariance structure. The rates of less than moderate to severe regret will be compared between groups at 6-months using a one-sided test about the appropriate contrast of model estimates.

SECONDARY OUTCOMES:
Quality of Life (EORTC QLQ-C30) | Up to 6 months
  Will compare QOL measures based on the European Organization for Research and Treatment of Cancer Core Quality of Life Questionnaire (EORTC QLQ-C30) between the provision of QOL information versus usual care for standard of care surgery or SBRT treatment.
Quality of Life (QOL) | Up to 6 months
  Will compare QOL measures based on the lung cancer- specific questionnaire (EORTC QLQ-LC13) between the provision of QOL information versus usual care for standard of care surgery or SBRT treatment.
Difference in consideration of regret | Up to 6 months
  Compare decisions about treatment for early stage lung cancer and examined whether regret is a consideration in treatment decisions between those who received the quality of life fact sheet and those who did not.

CONTACTS AND LOCATIONS:
Overall Officials: Anurag K Singh, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States